CLINICAL TRIAL: NCT00133835
Title: Comparison of ESWL Alone and ESWL Combined With Endoscopic Drainage of the Main Pancreatic Duct for Painful Chronic Pancreatitis
Brief Title: Comparison of ESWL Alone and ESWL + Endoscopy for Painful Chronic Pancreatitis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Erasme University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 97.187
Record Dates: First submitted 2005-08-22; First posted 2005-08-24 (Estimated); Last update posted 2022-03-09 (Actual); Status verified 2005-07

CONDITIONS: Pancreatitis
Keywords: Randomized controlled trial; Lithotripsy; Cholangiopancreatography, Endoscopic Retrograde; Abdominal pain
MeSH Terms: conditions — Pancreatitis; Abdominal Pain | interventions — Lithotripsy

INTERVENTIONS:
Procedure: Extracorporeal shock wave lithotripsy
Procedure: Endoscopic drainage of the main pancreatic duct

SUMMARY:
Endoscopy is an established method of treatment for painful obstructive calcified pancreatitis. It involves the disintegration of calcifications using extracorporeal shock wave lithotripsy (ESWL) followed by endoscopic removal of stone fragments possibly associated with stent insertion. A pilot study suggests that ESWL alone relieves pain in calcified chronic pancreatitis (CP). The aim of this study is to compare both techniques in a randomized controlled trial.

DETAILED DESCRIPTION:
Endoscopic drainage of the main pancreatic duct is an established method of treatment of painful obstructive calcified chronic pancreatitis (CP). It involves disintegration of calcifications using extracorporeal shock wave lithotripsy (ESWL) followed by endoscopic removal of stone fragments, possibly associated with stent insertion. A pilot study suggests that ESWL alone in calcified CP is followed by spontaneous elimination of stone fragments and pain relief, without sphincterotomy. After ESWL alone, the exocrine function was found to return to normal values in some cases. Potential benefits include lower costs and morbidity as well as wider availability compared to endoscopic techniques.

The primary outcome of this randomized controlled trial is to compare the relapse of pain at 2 years after treatment with ESWL alone or endoscopic treatment, consisting of ESWL followed by endoscopic stone extraction. Secondary outcomes include a comparison of technical results (as assessed by abdominal CT Scan 1 week after the last intervention and secretin-enhanced magnetic resonance at 1 month), complication rates, and treatment-related costs in both groups.

Patients are eligible to participate in the study according to the following criteria:

Inclusion criteria :

* painful chronic pancreatitis (abdominal pain attack during the preceding 12 months);
* at least 1 calcified stone greater than 4 mm in one of its axes in the cephalic or corporeal portion of the main pancreatic duct with upstream duct dilation;
* written informed consent obtained from the patient.

Exclusion criteria:

* history of treatment of the pancreas using ESWL, endoscopy, or surgery;
* pancreatic collection greater than 2 cm in diameter at magnetic resonance or CT Scan;
* alkaline phosphatase levels greater than twice the upper limit of normal values or signs of cholangitis;
* age below 18 years;
* pregnancy or lactation.

Pretherapeutic work-up will include detailed medical history (including date of the first episode of typical abdominal pain, date of diagnosis of CP, number of episodes of pain during the last year, alcohol intake, pain continuous or intermittent during the last episode, medication, intensity of the last episode of pain on a 10-point scale as previously described), blood chemistry, stool sampling (for elastase measurement), triolein breath test, plain abdominal film taken in four classical positions (left anterior oblique, right anterior oblique, lateral, and supine), CT Scan without contrast medium injection, and secretin-enhanced magnetic resonance cholangiopancreatography (S-MRCP).

After informed consent of the referring physician has been obtained, patients will be asked to participate in the study. If the patient accepts, after oral and written consent, he (or she) will be randomized to the ESWL or endoscopy group by opening an opaque sealed envelope numbered according to a table of random numbers.

ESWL will be performed in all patients using a electromagnetic lithotriptor as previously described. Shock-waves will be focused on the obstructing stones (if multiple stones are present, those responsible for MPD obstruction will be identified by comparing plain abdominal film, CT Scan and S-MRCP). ESWL sessions will be repeated if necessary, until stone fragmentation is obtained, as confirmed by abdominal plain film centered on the targeted area of the pancreas. At this time, treatment will be considered terminated in the ESWL group, patients in the endoscopy group will undergo endoscopy immediately, for endoscopic extraction of stone fragments possibly associated to stent insertion according to previously published criteria and techniques.

Cross-over: in the ESWL group, if no elimination of the fragments is observed one week after the last ESWL, endoscopic drainage of the main pancreatic duct will be carried out at this time in case of continuous pain. For patients without continuous pain, delayed spontaneous elimination of the fragments will be sought by CT Scan and S-MRCP 2 months after the last ESWL. Endoscopic drainage of the main pancreatic duct will be proposed during follow-up only to the patients presenting a painful attack of CP.

Follow-up will consist of clinical examination 1 month after treatment and every 6 months thereafter. Data collected will include pain relapses, ESWL, endoscopic and surgical procedures, weight change, plus any other seemingly unrelated medical treatments. In addition to this, a S-MRCP will be performed 1 month after treatment. Triolein breath test will be performed at 1 month and 1 year. Sampling of stools (for elastase measurement) will be obtained every year.

Costs will be calculated starting on the day of first treatment as previously described. Costs not directly related to the treatment of pain or of procedure-related complications (e.g., diabetes) will be disregarded.

ELIGIBILITY:
Inclusion Criteria:

* Painful chronic pancreatitis (>1 abdominal pain attack during the preceding 12 months)
* At least 1 calcified stone greater than 4 mm in one of its axes in the cephalic or corporeal portion of the main pancreatic duct (MPD) with upstream duct dilation
* Written informed consent obtained from the patient

Exclusion Criteria:

* History of treatment of the pancreas using ESWL, endoscopy, or surgery
* Pancreatic collection greater than 2 cm in diameter at magnetic resonance or CT scan
* Alkaline phosphatase levels greater than twice the upper limit of normal values or signs of cholangitis
* Age below 18 years
* Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 1998-03; Primary Completion 2022-02-21 (Actual); Study Completion 2022-02-21 (Actual)

PRIMARY OUTCOMES:
Relapse of pain at 2 years

SECONDARY OUTCOMES:
Diameter of the main pancreatic duct at 1 month
Complication rate at 1 month
Treatment-related costs of initial intervention and during follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marc Dumonceau, Principal Investigator — University Hospital, Geneva; Jacques Devière, Principal Investigator — Erasme University Hospital; Guido Costamagna, Principal Investigator — Catholic University of Roma
Locations (2):
- Department of Gastroenterology and Hepatopancretology; Erasme University Hospital, Brussels, Belgium
- Digestive Endoscopy Unit, Department of Surgery, Catholic University, Rome, Italy